CLINICAL TRIAL: NCT02877628
Title: Immunosuppressive Therapy Optimization: Development of a Population Pharmacokinetic-pharmacodynamic (PK-PD) Model in Liver Transplantation
Acronym: OPTILTH
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC13_8962_OPTILTH
Record Dates: First submitted 2016-08-16; First posted 2016-08-24 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Liver Transplantation
Keywords: pharmacokinetic; pharmacodynamic; tacrolimus; CYP3A5; liver transplantation
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Pharmacokinetic-pharmacodynamic model in liver transplantation — Biological: tacrolimus and calcineurin dosage, donor and recipient CYP3A5 and ABCB1 genotypes determination

SUMMARY:
Prospective, non-randomized, open Pharmacokinetic-Pharmacogenetic-Pharmacodynamic monocentric study. Donor and recipient CYP3A5 genotype and recipient ABCB1 will not be communicate to clinicians or patients during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18
* Liver transplant recipients
* Treated with an immunosuppressive protocol with tacrolimus
* Informed on the study and who did not refuse to participate

Exclusion Criteria:

* Patients who participate in a study with procedures incompatible with the present study.
* Patients with legal protection/deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with liver tranplantation
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-10-31 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Prediction of calcineurin inhibition, responsible for the immunosuppressive effect | Week 24
  Assessement of the relationships between tacrolimus dosage, whole-blood and intracellular concentrations
Prediction of calcineurin inhibition, responsible for the immunosuppressive effect | Week 24
  Assessement of the relationships between intracellular concentrations of tacrolimus and calcineurin activity
Prediction of calcineurin inhibition, responsible for the immunosuppressive effect | Week 24
  Assessement of the relationships between donor and recipient CYP3A5 and ABCB1 genotypes and dose/concentration of tacrolimus
Prediction of calcineurin inhibition, responsible for the immunosuppressive effect | Week 24
  Assessement of the relationships between intracellular concentration of tacrolimus and/or calcineurin activity and ACR, in patients treated with immediate release or modified-release formulation of tacrolimus

SECONDARY OUTCOMES:
Study of impact of pharmacogenetic and demographic data on tacrolimus intracellular concentration | Week 24
Evaluation of the role of the measurement of intracellular concentration as a longitudinal biomarker in preventing acute cellular graft (ACR) | Week 24
Study of variability of tacrolimus intracellular concentration according to its pharmaceutic form (immediate or sustained release) | Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France